CLINICAL TRIAL: NCT06635616
Title: Emergency Department Hypertension Management: Effects of Routine Oral Antihypertensive Agents on Emergency Management of Hypertension
Brief Title: Hypertension Management in Terms of Routine Agents
Status: Not yet recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Etimesgut Military Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: hypertension
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Hypertension; Emergency Medicine
Keywords: hypertension; emergency medicine; oral antihypertensive agents
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- diuretics: patients prescribed diuretics for oral treatment admitted to emergency service with elevated blood pressure
- Beta Blockers: patients prescribed Beta Blockers for oral treatment admitted to emergency service with elevated blood pressure
- Calcium Channel Blockers: patients prescribed Calcium Channel Blockers for oral treatment admitted to emergency service with elevated blood pressure
- ACE (angiotensin converting enzyme) Inhibitors: patients prescribed ACE (angiotensin converting enzyme) Inhibitors for oral treatment admitted to emergency service with elevated blood pressure
- ARB( angiotensin receptor blockers): patients prescribed ARB( angiotensin receptor blockers) for oral treatment admitted to emergency service with elevated blood pressure
- combination: patients prescribed combination agents for oral treatment admitted to emergency service with elevated blood pressure

SUMMARY:
known hypertensive patients admitted to emergency department with increased blood pressure will be evaluated in terms of antihypertensive agents given at hospital, degree of blood pressure decrease, hospital stay and laboratory and imaging tests ordered. The impact of routine oral antihypertensive agents used by the patients on these parameter will be assessed.

DETAILED DESCRIPTION:
Hypertensive patients account for approximately 1-25% of annual emergency department visits . While this figure varies by region, hypertensive patients are among the groups that contribute significantly to emergency department crowding and workload . Hypertensive emergencies constitute about 0.3-0.9% of all patients, and this number is rapidly increasing each year .

The 2017 AHA hypertension guidelines emphasize that severe elevations in blood pressure (hypertensive crisis and hypertensive urgency) do not require emergency department visits or referrals unless there is end-organ damage . It is noted that treatment in these patients typically involves dose adjustment or a change in medication .

The 2023 ESC hypertension guidelines recommend that in patients presenting to the emergency department with a hypertensive crisis, blood pressure should be gradually lowered with oral agents over a 24-48 hour period. These patients do not usually require hospital admission but can be monitored in an outpatient setting for clinical evaluation. It is noted that their blood pressure may remain elevated upon discharge from the emergency department, and follow-up in a clinic is necessary for reevaluation of chronic therapy .

Some studies have indicated that both oral and intravenous treatments are preferred for patients presenting with hypertensive crises, highlighting that the approach can vary from physician to physician .

When evaluating literature reviews, published guidelines, and conducted studies, it is observed that there are differences between European and American approaches in defining and treating hypertensive crisis, as well as variability in physician management of these patients .

In our study, we plan to evaluate the effect of emergency department treatment on lowering blood pressure in known hypertensive patients (≥140/80) without end-organ damage. Additionally, we aim to assess the impact of the antihypertensive agents that patients routinely use on their length of stay in the emergency department, as well as the frequency and effectiveness of the medications used, and the target blood pressure values achieved post-treatment according to guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 and older.
2. Blood pressure measured at ≥140/80.
3. Diagnosis of essential hypertension.

Exclusion Criteria:

1. Pregnant patients.
2. Individuals without a prior diagnosis of hypertension.
3. Patients with end-organ damage (hypertensive emergency).
4. Patients whose routine antihypertensive agents are unavailable.
5. Patients who leave the clinic without permission, making follow-up data inaccessible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with known hypertension admitted to emergency department with elevated blood pressure
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
routine use of oral antihypertensive agents and its effects on emergency service care | from enrollment to the end of follow up duration of 7 days
  emergency service blood pressure target achievement duration changes depending on routine oral antihypertensive agent prescribed

CONTACTS AND LOCATIONS:
Overall Officials: Elif HAMZACEBIOGLU KAYISOGLU, Specialist, Study Director — Etimesgut Military Hospital; Gulsen AKCAY, Ass. Prof., Principal Investigator — Ankara Etlik City Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Etlik City Hospital, Ankara
  - Etimesgut Military Hospital, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salvetti M, Paini A, Colonetti E, Tarozzi L, Bertacchini F, Aggiusti C, Stassaldi D, Rosei CA, Rosei EA, Muiesan ML. Hypertensive emergencies and urgencies: a single-centre experience in Northern Italy 2008-2015. J Hypertens. 2020 Jan;38(1):52-58. doi: 10.1097/HJH.0000000000002213. PMID 31415308
- [Background] Nowicki J, Silka W, Zalustowicz A, Rajzer M, Olszanecka A. Uncontrolled hypertension and hypertensive urgency: One-year single-center emergency department experience. Kardiol Pol. 2024;82(4):407-415. doi: 10.33963/v.phj.100025. Epub 2024 Apr 12. PMID 38606743
- [Background] Astarita A, Covella M, Vallelonga F, Cesareo M, Totaro S, Ventre L, Apra F, Veglio F, Milan A. Hypertensive emergencies and urgencies in emergency departments: a systematic review and meta-analysis. J Hypertens. 2020 Jul;38(7):1203-1210. doi: 10.1097/HJH.0000000000002372. PMID 32510905